CLINICAL TRIAL: NCT02005549
Title: A Phase II Study of Bevacizumab With Docetaxel and Capecitabine in the Neoadjuvant Setting for Breast Cancer Patients
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Chemotherapy in Patients With Primary Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19869
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel; Capecitabine

ARMS (1):
- Neoadjuvant Therapy (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: docetaxel; Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15 mg/kg iv on Day 1 of each 3-week cycle, 5 cycles
Drug: docetaxel — 75 mg/m2 on Day 1 of each 3-week cycle, 6 cycles
Drug: capecitabine [Xeloda] — 950 mg/m2, orally twice daily, evening of Day 1 until morning of Day 15, followed by a 7 day rest period, every 3 weeks

SUMMARY:
This study will evaluate the effect of Avastin (15mg/kg iv) in combination with Docetaxel and Xeloda, given as pre-operative therapy to patients with primary breast cancer. Avastin will be administered every 3 weeks, for the first 5 cycles of chemotherapy. The anticipated time on study treatment is 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* female patients, 18-70years of age;
* histologically-proven invasive breast cancer;
* no prior or current neoplasm except for non-melanoma skin cancer, or in situ cancer of the cervix;
* no distant disease/secondary cancer.

Exclusion Criteria:

* pregnant or lactating women;
* pre-operative local treatment for breast cancer;
* prior or concurrent systemic antitumor therapy;
* clinically significant cardiac disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (1):
- Salzburg, Austria

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab+Docetaxel+Capecitabine: Participants received bevacizumab, 15 milligrams/kilogram (mg/kg) intravenously (IV), followed by docetaxel 75 mg per square meter (mg/m^2) IV on Day 1 and capecitabine 950 mg/m^2 orally (PO) twice daily (BID) within 30 minutes after the end of a meal, starting the evening of Day 1 and continuing until the morning of Day 15 (followed by a 7-day rest period) for a maximum of five 3-week cycles.
Period: Overall Study
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population. All participants who received at least one dose of study drug.
Groups:
- Bevacizumab+Docetaxel+Capecitabine: Participants received bevacizumab, 15 mg/kg IV, followed by docetaxel 75 mg/m^2 IV on Day 1 and capecitabine 950 mg/m^2 PO BID within 30 minutes after the end of a meal, starting the evening of Day 1 and continuing until the morning of Day 15 (followed by a 7-day rest period) for a maximum of five 3-week cycles.
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 48 [34 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Response (pCR)
Description: pCR was defined as the absence of signs for invasive tumor in the final surgical sample as judged by the local pathologist. Surgery was performed 2 to 4 weeks after the last chemotherapy cycle.
Time Frame: Baseline, 20-24 weeks (final surgery, performed 2 to 4 weeks after the last chemotherapy cycle [Week 18])
Population: ITT population; participants evaluable for response included those participants who received a minimum of 3 cycles of treatment (9 weeks on study) with final surgery performed and the samples and reports available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Number analyzed (Participants) | 18
percentage of participants | 22.22 [6.41 to 47.64]

2. Secondary Outcome: Percentage of Participants With pCR, Clinical Complete Response (CR), or Clinical Partial Response (PR)
Description: Percentage of participants with pCR plus the percentage of participants without pCR who achieved CR or PR as measured by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal (short axis less than [<] 10 millimeters [mm]). No new lesions. PR was defined as greater than or equal to (≥) 30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, 20-24 weeks (final surgery, performed 2 to 4 weeks after the last chemotherapy cycle [Week 18])
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Number analyzed (Participants) | 18
percentage of participants | 72.22 [46.52 to 90.31]

3. Secondary Outcome: Percentage of Participants Undergoing Breast-Conserving Surgery
Description: Percentage of participants undergoing a breast-conserving procedure versus a modified radical mastectomy at final surgery, performed 2 to 4 weeks after the last chemotherapy cycle (Week 18)
Time Frame: 20-24 weeks (final surgery, performed 2 to 4 weeks after the last chemotherapy cycle [Week 18])
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Number analyzed (Participants) | 18
percentage of participants | 83 [59 to 96]

ADVERSE EVENTS:
Time Frame: Baseline, every three weeks (Cycles 1 through 6), end-of-treatment, to 28 days after last dosage of study drug.
Description: An adverse event is any undesirable event associated with the use of a drug, whether or not considered drug related, and includes any side effect, injury, toxicity, or sensitivity reactions. It also includes any undesirable clinical or laboratory event which is not normally observed in the participant.
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Serious Adverse Events (participants affected / at risk) | 5/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Docetaxel+Capecitabine (N=18)
Deep vein thrombosis (Vascular disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Impaired healing (General disorders) | 1
Neutropenic infection (Infections and infestations) | 1
Contralateral breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Docetaxel+Capecitabine (N=18)
Alopecia (Skin and subcutaneous tissue disorders) | 17
Nail disorder (Skin and subcutaneous tissue disorders) | 12
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 8
Anaemia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Blood lactate dehydrogenase increased (Investigations) | 8
Weight decreased (Investigations) | 5
Alanine aminotransferased increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Pulse abnormal (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2
Fatigue (General disorders) | 6
Asthenia (General disorders) | 1
General physical health deterioration (General disorders) | 1
Impaired healing (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Dysgeusia (Nervous system disorders) | 4
Polyneuropathy (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Rhinitis (Infections and infestations) | 3
Laryngitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Neutropenic infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Hot flush (Vascular disorders) | 3
Deep vein thrombosis (Vascular disorders) | 2
Thrombophlebitis (Vascular disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Conjunctivitis (Eye disorders) | 2
Visual acuity reduced (Eye disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Procedural pain (Injury, poisoning and procedural complications) | 1
Wound complications (Injury, poisoning and procedural complications) | 1
Contralateral breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

LIMITATIONS AND CAVEATS:
Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.